CLINICAL TRIAL: NCT02927392
Title: The Impact of Estrogen Status on the Biological Function of Brown Adipose Tissue in Women Measured Using Quantitative PET/CT
Brief Title: Brown Adipose Tissue Activity in Pre- and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Ottawa (Other); Université de Sherbrooke (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1479; 1R01DK112260-01 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-07 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Menopause; Obesity
MeSH Terms: conditions — Obesity | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-menopausal women (Experimental): To determine if natural declines in endogenous E2 contribute to changes in BAT activity, the investigators will compare BAT activity in pre-and post-menopausal women. We will also explore whether suppression of ovarian hormones in pre-menopausal women (using leuprolide acetate) impairs BAT activity.
  Interventions: Drug: Leuprolide acetate
- Post-menopausal women (No Intervention): To determine if natural declines in endogenous E2 contribute to changes in BAT activity, the investigators will compare BAT activity in pre-and post-menopausal women.

INTERVENTIONS:
Drug: Leuprolide acetate — A subset of premenopausal women will receive GnRHAG (leuprolide acetate) 3.75 mg/mo by intramuscular injection every 4 weeks for 24 weeks (6 doses).
  Other Names: Lupron
  Arms: Pre-menopausal women

SUMMARY:
The physiological relevance of brown adipose tissue (BAT) in humans is largely unknown. The investigators have shown that suppressing ovarian function in premenopausal women reduces resting energy expenditure (REE), and this is prevented by adding back estradiol (E2). The investigators preliminary data suggest that this may be due, in part, to reduced brown adipose tissue (BAT) activity. The overarching hypothesis is that BAT activity in humans is modulated by E2. To determine if natural declines in endogenous E2 contribute to changes in BAT activity, we will compare BAT activity in pre-and post-menopausal women. The investigators will also explore whether suppression of ovarian hormones in pre-menopausal women impairs BAT activity. BAT activity will be quantified using dynamic positron emission topography/computed tomography (PET/CT) imaging combined with 11C-acetate tracers. We will assess the thermogenic response of BAT by measuring cold-induced changes in REE, shivering, and skin and core temperature.

DETAILED DESCRIPTION:
Participants will be asked to perform studies to measure resting metabolic rate and activity of brown adipose tissue or brown fat. Brown fat is different from regular "white fat" in that it produces heat and burns calories. The investigators will measure how active brown fat is at normal room temperature and after participants have been exposed to cold.

The study will last 5-6 hours. It will consist of measurements made in warm temperatures and then after a period of cold exposure. For the cold exposure part of the study, participants will be asked to wear a cooling suit for 3 hrs. Skin temperature is normally about 90º Fahrenheit. The cooling suit will adjust the water temperature until your skin temperature is about 82º Fahrenheit. The suit will cover the entire body except for the face, hands, and feet. Participants may feel cold while wearing the suit and you may shiver some, but based on past studies, any shivering should be minor.

Before and after the cooling suit is turned on, body scans will be performed using a procedure called positron emission tomography (PET). These scans do not use radiation. Before the PET scans, the investigators will infuse radioactive tracer into an arm. These tracers have a low dose of radiation and will show us where the brown fat is and how active it is. One PET scan will be performed at room temperature, and the second scan will be performed after the cooling suit has been worn for 3 hours. Two additional scans using computed tomography (CT) will be performed at end of the study. CT scans are like an x-ray, and use radiation. The radiation dose in the CT scan is much higher than the tracers. When the CT scans are combined with the PET scans, we can separate brown fat from white fat.

15 pre-menopausal women will be asked to volunteer for a follow up study. For 5 months, pre-menopausal women in this study will receive monthly injections that contain a study drug (leuprolide) that reduces estrogen to postmenopausal levels. This drug is approved by the FDA to reduce estrogen for the treatment of uterine fibroids and endometriosis, but is not approved for use in healthy women. In this study, the drug is being used to decrease hormones to determine if this reduces brown fat activity. 6 months after the first injection, these women will be asked to repeat the PET/CT studies.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal volunteers will be healthy, eumenorrheic women, aged 18-45 yrs. Eumenorrheic status will be verified by regular menses (no missed cycles in previous year; cycle length 25-35 d).
* Postmenopausal volunteers will be healthy women who have no menses for at least 12 months

Exclusion Criteria:

- Body mass index (BMI) > 35 kg/m2

Additional exclusion criteria for premenopausal women

* Hormonal contraceptive use (past 6 mo.)
* Pregnant, lactating or intention to become pregnant during the period of study

Additional exclusion criteria for postmenopausal women

* History or current use of hormonal replacement therapy (HRT)
* Women who have undergone surgical menopause.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melanson, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Started | 44 | 25
Completed | 28 | 25
Not Completed | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-menopausal Women | Post-menopausal Women | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 15 | 43
  >=65 years | 0 | 10 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9) | 64 (8) | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 20 | 42
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Brown Adipose Tissue Volume
Description: Brown adipose tissue volume will be measured using the radioactive tracer 18Fluro-deoxyglucose.
Time Frame: 5-6 hrs
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Number analyzed (Participants) | 28 | 25
mL | 53.1 (42.5) | 20.6 (29.7)

2. Primary Outcome: Brown Adipose Tissue Activity -Warm Exposure
Description: Brown adipose tissue activity in warm temperatures will be measured using the radioactive tracer 11C-acetate
Time Frame: 5-6 hrs
Measure: Mean (Standard Deviation); unit: disintegration per min (dpm)
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Number analyzed (Participants) | 26 | 25
disintegration per min (dpm) | .557 (0.309) | .631 (.283)
Statistical Analysis 1: Comparison: Pre-menopausal Women vs Post-menopausal Women; Test type: Other; p < 0.0001, ANOVA

3. Primary Outcome: Brown Adipose Tissue Activity - ColdExposure
Description: Brown adipose tissue activity after cold exposure will be measured using the radioactive tracer 11C-acetate
Time Frame: 5-6 hrs
Measure: Mean (Standard Deviation); unit: disintegration per minute (dpm)
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Number analyzed (Participants) | 27 | 25
disintegration per minute (dpm) | 1.277 (.851) | .906 (.544)

4. Secondary Outcome: Resting Energy Expenditure - Before Cold Exposure
Description: Resting energy expenditure is the calories burned when a person is at rest.
Time Frame: 5-6 hrs.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Number analyzed (Participants) | 28 | 25
kcal/day | 1334 (205) | 1223 (189)

5. Secondary Outcome: Resting Energy Expenditure - After Cold Exposure
Description: Resting energy expenditure is the calories burned when a person is at rest.
Time Frame: 5-6 hrs
Measure: Mean (Standard Deviation); unit: kcal/h
Arm/Group | Pre-menopausal Women | Post-menopausal Women
Number analyzed (Participants) | 28 | 25
kcal/h | 93.6 (25.3) | 85.0 (19.3)

ADVERSE EVENTS:
Time Frame: For participants in the cross-sectional study, the period of time they were in the study was 1-3 months. For premenopausal women who completed the suppression study, they period of time they were in the study was 7-8 months.
Arm/Group | Pre-menopausal Women | Post-menopausal Women
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02927392/Prot_SAP_000.pdf